CLINICAL TRIAL: NCT01025609
Title: Dietary Patterns & There Relationship to Cardiovascular Disease Risk Factors In Individuals With Chronic Spinal Cord Injury
Brief Title: Dietary Patterns and Cardiovascular (CVD) Risk in Spinal Cord Injury (SCI) Factors In Individuals With Chronic Spinal Cord Injury
Acronym: SCIDS
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 04-09-17E
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2022-06-29 (Actual); Status verified 2021-07

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; cardiovascular disease; dietary patterns
MeSH Terms: conditions — Spinal Cord Injuries; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will look at dietary patterns in individuals with chronic spinal cord injuries and the relationship between these dietary patterns and cardiovascular disease risk factors. The study is a supplement to the Coronary Artery Risk Development in Young Adults (CARDIA) study. The dietary history from CARDIA will be used. The investigators' primary hypothesis is the following: Greater whole-grain and dietary fiber intake will be favorably associated with adiposity (BMI and WC) and metabolic CVD risk factors (fasting glucose, fasting insulin, HOMA-IR, diabetes, hsCRP, TC, HDL-C, triglycerides, TC/HDL-C ratio, non-HDL-C, and systolic and diastolic blood-pressure) among a sample of individuals with SCI aged 38-50 who have been injured >1 year.

DETAILED DESCRIPTION:
This study is a cross-sectional study. It will look at dietary patterns in individuals with chronic spinal cord injuries and the relationship between these dietary patterns and cardiovascular disease risk factors. The study is a supplement to the Coronary Artery Risk Development in Young Adults (CARDIA) study. The dietary history from CARDIA will be used. The investigators' primary hypothesis is the following: Greater whole-grain and dietary fiber intake will be favorably associated with adiposity (BMI and WC) and metabolic CVD risk factors (fasting glucose, fasting insulin, HOMA-IR, diabetes, hsCRP, TC, HDL-C, triglycerides, TC/HDL-C ratio, non-HDL-C, and systolic and diastolic blood-pressure) among a sample of individuals with SCI aged 38-50 who have been injured >1 year.

ELIGIBILITY:
Inclusion Criteria

* Male or female, black or white with SCI due to a nonvascular insult that caused an acute spinal cord injury (i.e. traumatic injury, transverse myelitis without a diagnosis of multiple sclerosis, surgical complication, or benign neoplasm) at least 1 year prior to enrollment including ASIA A,B,C
* Age at time of enrollment: > 38 years and <55 years (i.e., on or after 38th birthday and before 55th birthday)
* Voluntary, informed consent of participant
* Participant willing to comply with the testing protocols and questionnaires
* Communication and comprehension sufficient for compliance with all testing procedures and measures Exclusion Criteria
* SCI of a vascular or malignant etiology
* Pregnancy, end-stage renal disease, treatment for cancer except for non-melanoma skin cancer in the past five years
* Injury < 1 years prior to enrollment
* ASIA D
* Chronic, nontobacco substance-abuse

Ages: 38 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 100 individuals with chronic spinal cord injuries
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Whole-grain intake | Day - 30
  Average number of whole grain servings per day
Fruit and vegetable intake | Day - 30
  Average number of fruit and vegetable servings per day
Dairy intake | Day - 30
  Average number of dairy servings per day

SECONDARY OUTCOMES:
Waist circumference | Year 1
Total cholesterol | Year 1
HDL-C | Year 1
LDL-C | Year 1
Triglycerides | Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Shreiner, PhD, Principal Investigator — University of Minnesota; Jesse A. Lieberman, M.D., Study Director — Carolinas Rehabilitation/Carolinas Medical Center
Locations (1):
- Carolinas Rehabilitation, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lieberman J, Goff D Jr, Hammond F, Schreiner P, Norton HJ, Dulin M, Zhou X, Steffen L. Dietary intake and adherence to the 2010 Dietary Guidelines for Americans among individuals with chronic spinal cord injury: a pilot study. J Spinal Cord Med. 2014 Nov;37(6):751-7. doi: 10.1179/2045772313Y.0000000180. Epub 2014 Jan 3. PMID 24621049